CLINICAL TRIAL: NCT00056069
Title: Differences in Parental Caregiving Demands in Childhood Acute Lymphoblastic Leukemia by Length of Infusion Therapy
Brief Title: Study of the Physical and Emotional Needs of Parents Caring for Children Receiving Chemotherapy for Acute Lymphoblastic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCL01P3; COG-ACCL01P3 (Other: Children's Oncology Group); CDR0000271934 (Other: NCI); NCI-2012-02522 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U10CA095861 (NIH)
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Leukemia
Keywords: psychosocial effects of cancer and its treatment; childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Observational (Experimental): Questionnaire Administration: Participants complete questionnaires regarding caregiver demands and family information over 25-30 minutes within 3-4 months of the initiation of the child's treatment and at the completion of the first year of the child's treatment.
  Interventions: Other: questionnaire administration

INTERVENTIONS:
Other: questionnaire administration — Participants complete questionnaires regarding caregiver demands and family information over 25-30 minutes within 3-4 months of the initiation of the child's treatment and at the completion of the first year of the child's treatment.
  Other Names: Ancillary studies

SUMMARY:
RATIONALE: Studying the physical and emotional needs of parents who are caring for children receiving chemotherapy for cancer may help doctors plan effective treatments for the patient that allow for improved quality of life of the patient's family.

PURPOSE: This clinical trial is studying the different physical and emotional needs of parents whose children are undergoing chemotherapy for acute lymphoblastic leukemia either in an outpatient clinic or in the hospital.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the caregiving demands reported by parents of children with acute lymphoblastic leukemia receiving methotrexate on 2 different infusion schedules (inpatient care vs outpatient care).
* Compare the change in caregiving demands on these parents over time, in terms of physical and emotional care, the need to make family arrangements, the need to communicate about the child's care, the need to gather information about the child's health status, and the effect on family well-being.

OUTLINE: Participants complete questionnaires regarding caregiver demands and family information over 25-30 minutes within 3-4 months of the initiation of the child's treatment and at the completion of the first year of the child's treatment.

PROJECTED ACCRUAL: A total of 164 participants will be accrued for this study within 0.8 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Parent or legal guardian who is the primary caregiver of a patient enrolled on COG-P9904 or COG-P9905 protocol

  * Patient has not yet received week 13 of therapy

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Able to understand English

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2002-12; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Event Free Survival | Length of study

SECONDARY OUTCOMES:
Determine whether caregivers whose child is randomized to receive the 24-hour methotrexate infusion will report lower caregiving demand than will caregivers whose child is randomized to receive the 4-hour infusion | Length of study
Total score from the CMCC | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Diane Keegan Wells, RN, MSN, CPNP, Study Chair — University of Maryland Greenebaum Cancer Center
Locations (122):
- United States (107):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama Cancer Research Institute, Mobile, Alabama
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Stanford Cancer Center at Stanford University Medical Center, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Kaiser Foundation Hospital - San Diego, San Diego, California
  - Children's Hospital and Health Center - San Diego, San Diego, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Yale Comprehensive Cancer Center at Yale University School of Medicine, New Haven, Connecticut
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Joe DiMaggio Children's Hospital at Memorial, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Sacred Heart Children's Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Children's Hospital of Tampa, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Scottish Rite Campus, Atlanta, Georgia
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Pediatric Specialty Clinic at Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Walter Reed Army Medical Center, Silver Spring, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler Air Force Base, Keesler Air Force Base, Mississippi
  - University of Missouri - Columbia, Columbia, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Schneider Children's Hospital, New Hyde Park, New York
  - Mount Sinai Medical Center, New York, New York
  - Beth Israel Medical Center - Singer Division, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Leo W. Jenkins Cancer Center at Pitt County Memorial Hospital, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - East Tennessee State University Cancer Center at Johnson City Medical Center, Johnson City, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Children's Cancer Center and Hematology Service at Texas Children's Hospital, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MBCCOP - South Texas Pediatrics, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Center for Cancer Prevention and Care at Scott and White Clinic, Temple, Texas
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - INOVA Fairfax Hospital, Falls Church, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Carilion Medical Center for Children at Roanoke Community Hospital, Roanoke, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (3):
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
- Canada (8):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre de Recherche du Centre Hospitalier de l'Universite Laval, Sainte-Foy, Quebec
- University Medical Center Groningen, Groningen, Netherlands
- San Jorge Children's Hospital, Santurce, Puerto Rico
- Switzerland (2):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva